CLINICAL TRIAL: NCT01994681
Title: Testing Spectrosense EVA System for Detection of Pancreatic Cancer by Analyzing Volatile Organic Compounds (VOCs) in Exhaled Air
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rauscher, Gregory E., M.D. PA (Individual)
Collaborators: Spectrosense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 00004108
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Pancreatic Cancer
- Healthy

SUMMARY:
Volatile Organic Compounds (VOC) in human breath are captured and analyzed by the Spectrosense EVA system, which is combination of a gas chromatography (GC) and software algorithm. The objective is to obtain a set or sets of VOC bio-markers that will provide the best discrimination between Pancreatic Cancer sick population and healthy population. The gold standard for identifying sick/healthy population is biopsy proven Pancreatic cancer.

ELIGIBILITY:
Pancreatic cancer Group

Inclusion Criteria:

* Age from 18 years old
* Pancreatic cancer positive biopsy
* Before any treatment
* Signed Informed Patient Consent

Exclusion Criteria:

* Age under 18 years old
* Neoadjovant treatment
* Post surgery for Pancreatic cancer
* A history of any other cancer type, except skin cancer that is not melanoma

Healthy Group

Inclusion Criteria:

* Healthy patients
* No history of Pancreatic cancer
* Signed Informed Patient Consent

Exclusion Criteria:

* History of Pancreatic cancer
* Pancreatic cancer background in the family
* A history of any other cancer type, except skin cancer that is not melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cancer, biopsy confirmed, before treatment, ages above 18. vs. Healthy subjects without pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Obtaining a set or sets of VOC bio-markers that will provide the best discrimination between Pancreatic Cancer sick population and healthy population. | Baseline
  An optimization algorithm will select VOCs that will provide maximal sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gutierrez, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States